CLINICAL TRIAL: NCT01560845
Title: Autologous Bone Marrow Stem Cells Infusion Through Hepatic Artery in Open Abdominal Portal Hypertension Surgery for the Treatment of Liver Cirrhosis: a Prospective, Non-randomized, Controlled Study
Brief Title: ABMSC Infusion Through Hepatic Artery in Portal Hypertension Surgery for the Treatment of Liver Cirrhosis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Qiqiang Zeng, the secretary-general of stem cell research center of Wenzhou Medical College, Wenzhou Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WZMC1-10-1
Record Dates: First submitted 2012-03-18; First posted 2012-03-22 (Estimated); Last update posted 2012-03-22 (Estimated); Status verified 2012-03

CONDITIONS: Liver Cirrhosis; Portal Hypertension; Hepatic Decompensation; Surgery
Keywords: autologous bone marrow stem cells; portal hypertension; surgery; liver cirrhosis
MeSH Terms: conditions — Liver Cirrhosis; Hypertension, Portal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ABMSCi plus surgery group (Experimental): Autologous bone marrow stem cells infusion through hepatic artery in open abdominal portal hypertension surgery
  Interventions: Procedure: Autologous bone marrow stem cells infusion （ABMSCi） plus abdominal portal hypertension surgery
- portal hypertension surgery group (No Intervention): only portal hypertension surgery for this group patients
  Interventions: Procedure: open abdominal portal hypertension surgery

INTERVENTIONS:
Procedure: Autologous bone marrow stem cells infusion （ABMSCi） plus abdominal portal hypertension surgery — Immediately after the harvest of ABMSC, the modified Sugiura procedure was performed for the patients who were assigned to the study group. The time of ABMSC separation and purification was 2.5-3 hours which had to be completed before the conclusion of portal hypertension surgery (3-3.5 hours). ABMSC was infused into proper hepatic artery through right gastric artery during the portal hypertension surgery
  Arms: ABMSCi plus surgery group
Procedure: open abdominal portal hypertension surgery — the modified Sugiura procedure was performed for the patients
  Arms: portal hypertension surgery group

SUMMARY:
In recent years, the safety and efficacy of autologous bone marrow stem cells infusion (ABMSCi) therapy were confirmed. The investigators attempted to infuse autologous bone marrow stem cells (ABMSC) through inserting a catheter into right gastric artery as far as proper hepatic artery after finishing open abdominal portal hypertension surgery. The present study was designed to treat bleeding from esophageal varices and hypersplenism and hopefully to improve the liver function as well.

DETAILED DESCRIPTION:
1. ABMSC mobilization and harvest

   * For harvesting more ABMSC, ABMSC mobilization was induced by rhG-CSF (Gran○R), administered subcutaneously at a dose of 300μg daily for three consecutive days before open abdominal portal hypertension surgery.
   * Bone marrow (160-200ml) of the patients was harvested from both posterior superior iliac according to standard procedures under local anaesthesia and was collected in a plastic bag containing heparin.
2. Open abdominal portal hypertension surgery

   - Immediately after the harvest of ABMSC, the modified Sugiura procedure was performed for the patients who were assigned to the study group. The same surgical procedure was also performed for the control group (without harvest of ABMSC and ABMSC infusion).
3. ABMSC separation and infusion

   * While performing the portal hypertension surgery, ABMSC was separated and purified in a class 10,000 clean laboratory. After fat and bony particles were removed by filtration, collected cells were moved to a cell-processing device. We used the reagent kit ([Patent Number] ZL 2006 1 0106875.5; [Number of Criteria Applicable] YZB/NING YIN 0008-2008; [Researcher and Developer] Wealthlin Science & Technology Inc., Canada; [Producer] Ningxia Zhonglianda Biotech Co., Ltd.). The reagents adopt the method of negative cells collection. Take the cells which intended to remove as target cells, and carry out the removal step-by-step. On the basis of this method, red blood cells, blood platelets, blood plasma will be completely removed with part of white cells and lymphocytes being remarkably removed as well while all the stem cells / progenitor cells are being well retained.
   * The nucleated cell (white blood cell) count of final ABMSC was measured by an automated complete blood count instrument and flow cytometry analysis. The number of mononuclear cells was counted manually under a microscope by Wright-Giemsa stain method. CD34 positive cells were determined by flow cytometry analysis.
   * The time of ABMSC separation and purification was 2.5-3 hours which had to be completed before the conclusion of portal hypertension surgery (3-3.5 hours). ABMSC was added to 10 ml saline and well mixed by shaking the vial gently. Before incision closure, the right gastric artery or right gastroepiploic artery was selected and a catheter was inserted. The catheter was pushed to reach the proper hepatic artery. The diameter of the catheter is 1.4mm, it is thin enough to easily been inserted to right gastric artery or right gastroepiploic artery (central venous catheterization, REF product NO.ES-04218, Arrow International, Inc.). The mixture of saline and AMBC was infused into hepatic artery at uniform speed for about two minutes. The catheter was removed after the ABMSCi. The puncture point of the right gastric artery was repaired using blood vessel suture or transfixed.
4. Statistical analysis - Categorical data are presented as absolute values and percentages, whereas continuous data are summarized as mean and Standard Deviation. Statistical analysis was performed using t-test for paired or unpaired samples. Time courses of measurements of liver function parameters were analyzed by repeated-measures ANOVA. The analyses were performed using the SPSS 15.0 statistical package (SPSS Inc., Chicago, IL, USA). All statistical analyses were based on two-tailed hypothesis tests with a significance level of p< 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced liver cirrhosis after hepatitis B resulted in bleeding from esophageal varices and hypersplenism, and needed open abdominal portal hypertension surgery;
2. Endoscopy evidence of showing severe gastric and esophageal varices;
3. Severe hypersplenism （white blood cells (WBC) <3×109/L and platelet (PLT) <100×109/L）;
4. Active bone marrow hyperplasia showed by bone marrow biopsy before surgery;
5. Age between 18 and 60 years;
6. Plasma albumin <35g/L, or mild ascites;

Exclusion Criteria:

1. Enlisted for liver transplantation
2. Diagnosis of hepatocellular carcinoma or other cancers
3. Other severe medical disease, and acute infection.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2010-06; Primary Completion 2013-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Child-pugh score | 1 month after treament

SECONDARY OUTCOMES:
Incidence of complications | within the first week after treatment
  postoperative pyrexia, intraperitoneal hemorrhage, intraperitoneal infection, malignant tumors of liver and other systems
Mortality | 1week, 1 month, 3 month, 6 month, 1 year and 2 year
blood test (hypersplenism) | whinin 7 days before treatment, 1 week,1,3, 6 and 12 months after treatment
  PLT and WBC
liver volume calculated by CT | whinin 7 days before treatment, 1 month and a year after treatment
  estimation of liver volume using CT
Indocyanine green (ICG) retention (clearance) | whinin 7 days before treatment, 1 week,1,3, 6 and 12 months after treatment
blood biochemistry | whinin 7 days before treatment, 1 week,1,3, 6 and 12 months after treatment
  1. alanine aminotransferase
  2. aspartate aminotransferase
  3. total bilirubin
  4. direct bilirubin
  5. The total bile acid (TBA)
  6. serum cholinesterase (CHE)
  7. albumin
  8. prothrombin time (PT)
  9. international normalized ratio (INR)

CONTACTS AND LOCATIONS:
Overall Officials: qiyu zhang, MD, Study Chair — First Affiliated Hospital of Wenzhou Medical University
Locations (1):
- the First Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang, China

REFERENCES:
- [Background] am Esch JS, Schmelzle M, Furst G, Robson SC, Krieg A, Duhme C, Tustas RY, Alexander A, Klein HM, Topp SA, Bode JG, Haussinger D, Eisenberger CF, Knoefel WT. Infusion of CD133+ bone marrow-derived stem cells after selective portal vein embolization enhances functional hepatic reserves after extended right hepatectomy: a retrospective single-center study. Ann Surg. 2012 Jan;255(1):79-85. doi: 10.1097/SLA.0b013e31823d7d08. PMID 22156926
- [Background] Kim JK, Park YN, Kim JS, Park MS, Paik YH, Seok JY, Chung YE, Kim HO, Kim KS, Ahn SH, Kim DY, Kim MJ, Lee KS, Chon CY, Kim SJ, Terai S, Sakaida I, Han KH. Autologous bone marrow infusion activates the progenitor cell compartment in patients with advanced liver cirrhosis. Cell Transplant. 2010;19(10):1237-46. doi: 10.3727/096368910X506863. Epub 2010 Jun 3. PMID 20525430
- [Background] Peng L, Xie DY, Lin BL, Liu J, Zhu HP, Xie C, Zheng YB, Gao ZL. Autologous bone marrow mesenchymal stem cell transplantation in liver failure patients caused by hepatitis B: short-term and long-term outcomes. Hepatology. 2011 Sep 2;54(3):820-8. doi: 10.1002/hep.24434. Epub 2011 Jul 14. PMID 21608000
- [Background] Terai S, Ishikawa T, Omori K, Aoyama K, Marumoto Y, Urata Y, Yokoyama Y, Uchida K, Yamasaki T, Fujii Y, Okita K, Sakaida I. Improved liver function in patients with liver cirrhosis after autologous bone marrow cell infusion therapy. Stem Cells. 2006 Oct;24(10):2292-8. doi: 10.1634/stemcells.2005-0542. Epub 2006 Jun 15. PMID 16778155